CLINICAL TRIAL: NCT02354989
Title: Effect on Exercise Capacity of Fixed Rate Vs Rate RESPONSIve Pacing in Patients With Permanent AF and Left Ventricular Dysfunction Underwent Radiofrequency Atrioventricular Junction aBLation and bivEntricular Pacing (RESPONSIBLE Study)
Brief Title: Rate RESPONSIVe Pacing in Patients With Permanent AF Underwent AV Node ABLation and bivEntricular Pacing (RESPONSIBLE)
Acronym: RESPONSIBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RESPONSIBLE
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Left Ventricular Dysfunction; Atrial Fibrillation
MeSH Terms: conditions — Ventricular Dysfunction, Left; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RR on first (Active Comparator): Rate Response on first
  Interventions: Device: Rate Response on first (VVI biventricular pacing)
- RR off first (Active Comparator): Rate Response off first
  Interventions: Device: Rate Response off first (VVI biventricular pacing)

INTERVENTIONS:
Device: Rate Response on first (VVI biventricular pacing) — Rate Response function is turned on in the device. The patients performs a 6 minute walking test. After a week Rate Response function is turned off and the patient performs a second 6 minute walking test.
  Arms: RR on first
Device: Rate Response off first (VVI biventricular pacing) — Rate Response function is turned off in the device. The patients performs a 6 minute walking test. After a week Rate Response function is turned on and the patient performs a second 6 minute walking test.
  Arms: RR off first

SUMMARY:
The purpose of this study is to evaluate the effect on distance covered in a 6 minute walking test of Rate Responsive pacing in patients with permanent atrial fibrillation and reduced left ventricular ejection fraction treated with atrioventricular junction ablation and biventricular pacing.

DETAILED DESCRIPTION:
Patients with permanent atrial fibrillation and reduced left ventricular ejection fraction treated with atrioventricular junction ablation and biventricular pacing will be enrolled. Two 6' walking test (6WT), one during VVI 70/min biventricular pacing (RR off) and the other during VVIR 70-120/min biventricular pacing (RR on), will be performed one week apart; patients will be randomly and blindly assigned with a 1:1 ratio to group A (first 6WT RR off) or B (first 6WT RR on). The difference between the two tests will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Permanent, refractory atrial fibrillation treated with atrio-ventricular node ablation and biventricular pacing
* Left ventricular systolic dysfunction
* Ability to perform a 6-minute walking test
* Completion of the 18th year of age

Exclusion Criteria:

* Contraindications to 6 minute walking test
* IV NYHA Class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The distance covered during the 6-minute walking test | 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Palmisano, MD, Principal Investigator — Azienda Ospedaliera "Card. G. Panico" - Tricase
Locations (7):
- Italy (7):
  - Università Politecnica delle Marche, Ancona, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - AO Pugliese-Ciaccio, Catanzaro, Catanzaro
  - Azienda Ospedaliera "Card. G. Panico", Tricase, Lecce
  - Seconda Università Napoli - A.O. Monaldi, Naples, Naples
  - AOU "Maggiore della Carità", Novara, Novara
  - Ospedale San Filippo Neri, Roma, Roma